CLINICAL TRIAL: NCT05204108
Title: Evaluation of the Preoperative Detection of Muscle Invasion in Bladder Cancer with Contrast-enhanced Ultrasonography: a Prospective Study
Brief Title: Preoperative Detection of Muscle Invasion in Bladder Cancer with Contrast-enhanced Ultrasonography
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Qiyun Ou, Dr., Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: SYSEC-KY-KS-2021-321
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Bladder Cancer
Keywords: Bladder Cancer; Contrast-enhanced Ultrasonography
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Contrast-enhanced Ultrasonography: To evaluate the diagnostic accuracy of CEUS for the preoperative staging of bladder cancer, which would benefit the implementation of efficient therapeutic strategies.

SUMMARY:
To evaluate the diagnostic accuracy of CEUS for the preoperative staging of bladder cancer, which would benefit the implementation of efficient therapeutic strategies.

DETAILED DESCRIPTION:
Bladder cancer can be grouped into non-muscle invasive bladder cancer (NMIBC) and muscle invasive bladder cancers (MIBC), the latter displaying high aggressiveness, a high degree of malignancy, complicated treatment, high propensity to metastasis, and poor prognosis. Currently, the clinical feasibility and accuracy of preoperative detection of muscle invasion in bladder cancer with contrast-enhanced ultrasonography (CEUS) are unclear.

To evaluate the diagnostic accuracy of CEUS for the preoperative staging of bladder cancer, which would benefit the implementation of efficient therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* (a) eligible patients should be 18-year-old or older;
* (b) patients should have a histologically or cytologically confirmed diagnosis of primary bladder cancer;
* (c) patients should not have had any surgery, chemotherapy, immunotherapy, or any therapy before CEUS diagnosis.

Exclusion Criteria:

* (a) participants with confirmed to have no carcinoma of the bladder;
* (b) participants with previous pelvic surgery, who had undergone therapy, any bladder surgery, or had received chemotherapy, radiotherapy or immunotherapy;
* (c) participants diagnosed with tumor recurrence or metastasis; (d) participants who were allergic to ultrasound contrast agents or could not tolerate CEUS examination, for instance, with recent myocardial infarction, angina pectoris, cardiac insufficiency, severe cardiac arrhythmia, a right/left cardiac shunt, severe pulmonary hypertension, uncontrolled systemic hypertension, acute respiratory distress syndrome, or chronic obstructive pulmonary disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who have a histologically or cytologically confirmed diagnosis of primary bladder cancer
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection of Muscle Invasion in Bladder Cancer | within 3 minutes
  To evaluate the preoperative staging of bladder cancer，whether it is non-muscle invasive bladder cancer (NMIBC) or muscle invasive bladder cancers (MIBC)

CONTACTS AND LOCATIONS:
Overall Officials: Baoming Luo, master, Principal Investigator — Department of Ultrasound in Medicine, Sun Yat-sen Memorial Hospital, Sun Yat-sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No